CLINICAL TRIAL: NCT06666140
Title: Ultrasound Functional Analysis of the Diaphragm and Upper Digestive Tract in Patients with Congenital Diaphragmatic Hernia
Brief Title: Preliminary Study of Pediatric Diaphragmatic Elastography
Acronym: ECHODIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9420; 2024-A01627-40 (Other: ANSM)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: congenital diaphragmatic hernia; ultrasound elastography; Chronic respiratory diseases; pulmonary hypertension; hypoplasia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group HDC (Experimental): 40 children with diaphragmatic hernia with or without prosthesis (HDC)
  Interventions: Other: Ultrasonic elastography
- Control Group (Other): 40 children free of any diaphragmatic pathology
  Interventions: Other: Ultrasonic elastography

INTERVENTIONS:
Other: Ultrasonic elastography — The measurement of diaphragmatic stiffness by shear waves is performed with a high-frequency linear ultrasound probe, intercostally, during apneas lasting a few seconds.
  After quantitative diaphragm thickness measurements, the ultrasound probe positioning is unchanged and regions of interest are placed in the patient's diaphragm thickness as well as in the adjacent liver or spleen (baseline). A stiffness result is obtained in kPa.
  The elastography measurement extends the duration of the ultrasound scheduled as part of patient care by only 10 minutes.
  The examination is painless and non-invasive.

SUMMARY:
This diaphragmatic elastography study is a preliminary pilot study to have first values of diaphragmatic stiffness in patients with a history of diaphragmatic hernia and to estimate the difference in stiffness compared to a group of patients without a history of hernia.

The hypothesis is to be able to correlate the values found with the patients' symptomatology and thus to better monitor patients by a simple, accessible, painless and reproducible diagnostic tool, to better understand their evolution and even to be able to anticipate possible difficulties (reflux, respiratory disorders, scoliosis, etc.).

Ultrasound elastography is a recent and clinically recognized method that uses an ultrasound approach to determine tissue stiffness in a non-invasive way.

ELIGIBILITY:
Inclusion Criteria:

* Group HDC:
* Patient followed at the CCMR (centres de compétence maladies rares) HDC of the Strasbourg University Hospital
* Aged between 3 and 17 years old inclusive
* Indifferent Sex
* Subject affiliated to a social protection health insurance scheme or beneficiary of such a scheme
* Subject able to understand the objectives and risks of the research and to provide dated and signed informed consent
* Subject who has been informed of the results of the preliminary medical examination

Control group:

* Subject followed in pediatric surgery
* Aged between 3 and 17 years old inclusive
* Indifferent Sex
* Subject affiliated to a social protection health insurance scheme or beneficiary of such a scheme
* Subject able to understand the objectives and risks of the research and to provide dated and signed informed consent
* Subject who has been informed of the results of the preliminary medical examination

Exclusion Criteria:

* Group HDC:

  * Refusal
  * Language barrier
  * Diaphragmatic surgery within the last 3 months
  * Patient with a viral picture in progress at the time of examination (assessment by the investigator)
  * Patient treated with muscle relaxant
  * Inability to give the subject informed information (subject in an emergency situation, difficulties in understanding the subject, etc.)
  * Subject under safeguard of justice
  * Subject under guardianship or curatorship
  * Pregnant or breastfeeding woman

Control group:

* Patient without thoracic pathology
* Refusal
* Language barrier
* Diaphragmatic pathology
* Any myopathy
* History of surgery of the upper digestive tract (esophagus and/or gastric and/or duodenal)
* Patient on muscle relaxant
* Patient with a viral picture in progress at the time of examination (assessment by the investigator)
* Patient treated with muscle relaxant
* Inability to give the subject informed information (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship or curatorship
* Pregnant or breastfeeding woman

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
To estimate the difference in diaphragm stiffness between a group of children with a diaphragmatic hernia with or without a prosthesis and a group of children without any diaphragmatic pathology. | Baseline
  Diaphragmatic rigidity in ultrasound elastographic analysis: measurement of diaphragm stiffness in shear wave elastography, in apnea (measurement in kPa).

SECONDARY OUTCOMES:
To estimate the difference in diaphragm stiffness between a group of children with a diaphragmatic hernia with a prosthesis and a group of children with a diaphragmatic hernia without a prosthesis. | Baseline
  Bilateral measurements for each subject of the diaphragm performed in mode B, Intercostal analysis in mode B
To estimate the difference in diaphragm stiffness between a group of children with a diaphragmatic hernia with a prosthesis and a group of children with a diaphragmatic hernia without a prosthesis. | Baseline
  Bilateral measurements for each subject of the diaphragm made in elastography.
To estimate the difference in diaphragm stiffness between a group of children with a diaphragmatic hernia with a prosthesis and a group of children with a diaphragmatic hernia without a prosthesis. | Baseline
  Bilateral measurements for each subject of the diaphragm made in TM mode, Analysis in M mode (time-movement).
To evaluate the correlation between age and the different parameters measured by ultrasound (on the total population and then within the 3 groups: no hernia, hernia with plaque, hernia without plaque) | Baseline
  Collection of age and the various parameters measured by ultrasound (diaphragmatic thickness and rigidity).
To estimate the association between patient stiffness and symptomatology in HDC subjects. | Baseline
  Measurement of rigidity and collection of symptoms

OTHER OUTCOMES:
To estimate the association between the absence of the prosthesis and the symptomatology of patients in HDC subjects | Baseline
  Collection of the presence of a prosthesis and the various symptoms
To estimate the difference in diaphragmatic mobility between a group of children with a diaphragmatic hernia (with or without a prosthesis) and a group of children without a hernia | Baseline
  Measurement of diaphragmatic mobility in a group of children with a diaphragmatic hernia (with or without a prosthesis) and a group of children without a hernia
To estimate the difference in pyloric position between a group of children with a diaphragmatic hernia (with or without a prosthesis) and a group of children without a hernia | Baseline
  Evaluation of the position of the pyloric (in strict axial section passing through the hepatic hilum, pylora normally visible. Estimate its position in cm (cranio caudal) in relation to the hilum if not in place) in a group of children with a diaphragmatic hernia (with or without a prosthesis) and a group of children without a hernia

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle TALON, Professor, Principal Investigator
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No